CLINICAL TRIAL: NCT03838523
Title: Non-concealed Placebo Treatment for Menopausal Hot Flushes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Yvonne Nestoriuc, Clinical Professor, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1705-100
Record Dates: First submitted 2019-01-29; First posted 2019-02-12 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Intervention Model Description: Women with ≥5 daily moderate to severe hot flushes of at least moderate bother are assigned 1:1 to a 4-week OLP treatment or no treatment. To explore the duration and maintenance of placebo effects, participants in the OLP group are randomized a second time and divided into two subgroups who either discontinue (OLP 4wk) or continue the OLP treatment (OLP 8wk) for another 4 weeks.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, patients and clinicians are aware of group assignment. Assessors are blinded to group assignment of participants. To prevent the breaking of blinding, participants are requested to not communicate their group affiliation when they have questions about the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OLP group (Experimental): At baseline, patients are given an explanation about why placebos without deception might be effective.
  Women allocated to this group receive an 4-week Open Label Placebo treatment. After 4 weeks, they are randomized again to either continue or discontinue the OLP treatment for another 4 weeks.
  Interventions: Other: Open Label Placebo
- No-treatment group (No Intervention): At baseline, patients are given an explanation about why placebos without deception might be effective.
  Women assigned to the no-treatment group do not receive any treatment as part of the study.

INTERVENTIONS:
Other: Open Label Placebo — See group description
  Arms: OLP group

SUMMARY:
It has been long viewed that placebos cannot be administered in accordance with ethical values because deception is instrumental to the placebo effect. This notion has been shaken up by studies on open-label placebos, showing that placebos can lead to positive effects even though their inert nature is disclosed.

Beneficial effects of double-blind placebos were found to be high in hot flush trials.

The objective of the study is to determine whether an open-label placebo (OLP) treatment is efficacious in alleviating hot flushes and bother among peri- and postmenopausal women.

DETAILED DESCRIPTION:
Beneficial effects of double-blind placebos were found to be high in hot flush trials. Recent studies demonstrating the efficacy of placebos without concealment provide a possible way to administer placebos in accordance with ethical and clinical values.

The objective of the study is to determine whether an open-label placebo (OLP) treatment is efficacious in alleviating hot flushes and bother among peri- and postmenopausal women.

In this assessor-blinded, randomized-controlled trial, women with ≥5 daily moderate to severe hot flushes of at least moderate bother are assigned 1:1 to a 4-week OLP treatment or no treatment. Both groups are informed about study objectives including a briefing about the inert nature of placebo pills, why OLP might be effective and the importance of the control group. To explore the duration and maintenance of placebo effects, participants in the OLP group are randomized a second time and divided into two subgroups who either discontinue (OLP 4wk) or continue the OLP treatment (OLP 8wk) for another 4 weeks. All participants receive three study visits: at enrolment, baseline (1 week later), and at post-treatment. A fourth study visit is conducted at 8-week follow-up with the two subgroups OLP 4wk and OLP 8wk. Qualitative interviews about subjective experiences with the OLP treatment are conducted with n = 8 women.

This trial will contribute to the evaluation of OLP treatments in clinical practice and further our understanding about the magnitude of placebo effects in hot flush treatments.

ELIGIBILITY:
Inclusion Criteria:

* at least 5 moderate or severe hot flushes per day, including night time
* all hot flushes have at least moderate ratings of bother (sum score ≥ 16 on the bother subscale of the Hot Flush Rating Scale (HFRS) [41]
* fluency in German language
* participants are in menopausal transition (irregularities ≥ 60 days in the past year), or postmenopausal (cessation of menstruation ≥ 1 year) [42].

Exclusion Criteria:

* use of hormonal therapy to treat hot flushes within the last 6 weeks before enrolment
* use of herbal remedies to treat hot flushes within the last 6 weeks before enrolment
* intake of selective serotonin reuptake inhibitors (SSRIs) or serotonin-norepinephrine reuptake inhibitors (SNRI) within the last 6 weeks before enrolment
* previous oophorectomy
* severe physical or cognitive impairments which would constitute a barrier to give informed consent
* severe depression and anxiety (≥ 9 sum score or ≥ 5 depression or anxiety subscore on the Patient Health Questionnaire-4)
* medical conditions which might interact with menopausal hot flushes such as untreated hyperthyroidism, alcohol abuse (excluded when ≥4 on AUDIT-C) and cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Difference in hot flush composite score | 4 weeks
  The group difference between OLP and no-treatment regarding frequency x severity of hot flushes as assessed by a portable paper diary in which participants record number and severity of hot flushes in realtime
Bother by hot flushes | 4 weeks
  The group difference between OLP and no-treatment regarding bother by hot flushes as assessed by the Hot Flush Rating Scale (Hunter & Liao, 1995). A sum score is calculated which ranges from 3 to 30 with higher scores indicating larger bother by hot flushes.

SECONDARY OUTCOMES:
Hot flush frequency | 4 weeks
  The group difference between OLP and no-treatment regarding the frequency of hot flushes as assessed by the diary
Health-related quality of life | 4 weeks
  The group difference between OLP and no-treatment regarding health-related quality of life as assessed by the Women's Health Questionnaire (WHQ; Hunter, 1992; Shin & Shin, 2012). Using the 37-item version of the WHQ, 8 subscales are calculated: Depressed mood, somatic symptoms, memory/concentration, vasomotor symptoms, anxiety/fears, sexual behaviour, sleep problems, and attractiveness. Although part of the questionnaire, we will not analyze the menstrual symptoms scale given that most women in our sample would be post-menopausal. Higher scores indicate better quality of life (e.g., higher scores in sexual behavior indicate that loss of sexual interest and sexual dissatisfaction is not experienced). Scores for each subscale range from 0 (poor health status) to 100 (good health status).
Global improvement | 4 weeks
  The group difference between OLP and no-treatment regarding global improvement as assessed by the Patient Global Impression of Change (Geisser et al. 2010; Guttoso et al. 2003)
Number of responders at week 4 | 4 weeks
  The group difference between OLP and no-treatment regarding number of responders at week 4 (≥50% in hot flush frequency at 4 weeks from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Nestoriuc, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunter MS, Liao KL. A psychological analysis of menopausal hot flushes. Br J Clin Psychol. 1995 Nov;34(4):589-99. doi: 10.1111/j.2044-8260.1995.tb01493.x. PMID 8563666
- [Background] Geisser ME, Clauw DJ, Strand V, Gendreau MR, Palmer R, Williams DA. Contributions of change in clinical status parameters to Patient Global Impression of Change (PGIC) scores among persons with fibromyalgia treated with milnacipran. Pain. 2010 May;149(2):373-378. doi: 10.1016/j.pain.2010.02.043. Epub 2010 Mar 23. PMID 20332060
- [Background] Guttuso T Jr, Kurlan R, McDermott MP, Kieburtz K. Gabapentin's effects on hot flashes in postmenopausal women: a randomized controlled trial. Obstet Gynecol. 2003 Feb;101(2):337-45. doi: 10.1016/s0029-7844(02)02712-6. PMID 12576259
- [Background] Hunter, M. S. The women's health questionnaire: A measure of mid-aged women's perceptions of their emotional and physical health. Psychology & Health, 7(1), 45-54, 1992.
- [Background] Shin H, Shin HS. Measurement of quality of life in menopausal women: a systematic review. West J Nurs Res. 2012 Jun;34(4):475-503. doi: 10.1177/0193945911402848. Epub 2011 Mar 25. PMID 21441417
- [Derived] Pan Y, Meister R, Lowe B, Winkelmann A, Kaptchuk TJ, Buhling KJ, Nestoriuc Y. Non-concealed placebo treatment for menopausal hot flushes: Study protocol of a randomized-controlled trial. Trials. 2019 Aug 16;20(1):508. doi: 10.1186/s13063-019-3575-1. PMID 31420050